CLINICAL TRIAL: NCT04534894
Title: Single-center Clinical Study of Early Diagnosis of Diabetic Cardiomyopathy With Fluorescence Lifetime Imaging Microscopy (FLIM)
Brief Title: Single-center Clinical Study of Early Diagnosis of Diabetic Cardiomyopathy With FLIM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-20-015
Record Dates: First submitted 2020-08-19; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Diabetic Cardiomyopathies
Keywords: diabetic cardiomyopathy; fluorescence lifetime imaging microscopy; metabolism
MeSH Terms: conditions — Diabetic Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DM group and DCM group: DM group: type 2 diabetes with normal diastolic function DCM group: type 2 diabetes with diastolic dysfunction
  Interventions: Diagnostic Test: fluorescence lifetime imaging microscopy

INTERVENTIONS:
Diagnostic Test: fluorescence lifetime imaging microscopy — collect 2mL of venous blood and use fluorescence lifetime imaging microscopy to exam NADH fluorescence characteristics of it

SUMMARY:
Diabetic Cardiomyopathy (DCM) is disease of myocardial structure and function which is independent of hypertension, coronary heart disease, heart valve abnormalities, and other types of heart disease. DCM affects approximately 12% of diabetics and also appeared in some patients with well-controlled blood glucose. There is no specific and effective diagnostic method of DCM currently. Since it is well known that the dysfunction of myocardial metabolism caused by hyperglycemia and insulin resistance induces DCM, the method of evaluation of the metabolism will assist the diagnosis of DCM.

Nicotinamide adenine dinucleotide (phosphate) (NAD(P)H) is one of important coenzymes involved in biological metabolism. Fluorescence lifetime microscopy (FLIM) can detect the metabolic status based on the fluorescence characteristics of NAD(P)H. Previous studies have reported that NAD(P)H fluorescence lifetime can be used to assess the metabolic status of living cardiomyocytes cultured in vitro, and metabolism changes related to myocardial infarction and heart failure in rats. the investigators detected the metabolic status by label-free FLIM on the myocardial tissues and blood plasma in a rat model of type 2 diabetic cardiomyopathy, and found FLIM could provide valuable information about the myocardial metabolism by detecting the NAD(P)H fluorescence lifetime of blood plasma.

Recently, The investigators have explored the method of the FLIM in clinical study. The investigators used FLIM to compare the NAD(P)H fluorescence lifetime of blood plasma in healthy participants, type 2 diabetic patients with normal diastolic function and with diastolic dysfunction. The results showed that the NAD(P)H fluorescence life parameter of a2 was lower in type 2 diabetic patients with diastolic dysfunction (30.5±2.7%) than in healthy participants (41.5±4.8%) and type 2 diabetic patients with normal diastolic function (37.8±3.7%). Therefore, The investigators propose FLIM can provide valuable information about the myocardial metabolism, and it can be used as a non-invasive, label-free, and rapid screening method of diagnosis of DCM.

In this study, the investigators will recruit 243 patients with type 2 diabetes and divide them into two groups: normal diastolic function group (DM Group) and diastolic dysfunction group (DCM Group), based on the symptoms, laboratory examination and echocardiographic results. Then FLIM will be applied to detect the NAD(P)H fluorescence characteristics of venous blood of all patients. After that, the correlation between the parameters of diastolic function (E peak, E/E' ratio, left atrial volume, NT-proBNP) and the parameters of metabolism status (NAD(P)H fluorescence life parameter of a2 and the ratio of bound state/free state NAD(P)H) will be analyzed. This study will verify FLIM is helpful to diagnose DCM.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-80 years old;
2. Echocardiography showed that the cardiac structure was normal and the left ventricular ejection fraction was more than 50%;
3. patients with type 2 diabetes mellitus;
4. Body mass index (BMI) was 20-25 kg / m2 in male and 19-24 kg / m2 in female;
5. No other drugs except hypoglycemic drugs were taken in one month;
6. Sign informed consent form before entering this study.

Exclusion Criteria:

1. Patients with type 1 diabetes mellitus;
2. Patients with diabetic ketoacidosis in the past;
3. Patients with coronary heart disease or with myocardial ischemia indicated by ECG;
4. EGFR < 60ml / min / 1.73m2 in recent one month;
5. Chronic liver disease, or the levels of alanine aminotransferase and glutamic oxaloacetic transaminase were more than 3 times of the upper limit of the normal before enrollment;
6. Abnormal thyroid function;
7. Abnormal tumor index;
8. Dyslipidemia;
9. Pregnant and lactating women;
10. Allergy to contrast media.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetes patients, divided into two groups, based on the diastolic funciton
Sampling Method: Probability Sample
Enrollment: 243 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
fluorescence characteristics of NAD(P)H in venous blood by FLIM can assist early diagnosis of diabetic cardiomyopathy | 12 month
  (NAD(P)H fluorescence life parameter of a2 (%) in venous blood is lower in DCM patients than DM patients.
fluorescence characteristics of NAD(P)H in venous blood by FLIM can assist early diagnosis of diabetic cardiomyopathy | 12 month
  the ratio of bound state/free state NAD(P)H) (%) is lower in DCM patients than DM patients.

CONTACTS AND LOCATIONS:
Overall Officials: guangyu chen, doctor, Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rubler S, Dlugash J, Yuceoglu YZ, Kumral T, Branwood AW, Grishman A. New type of cardiomyopathy associated with diabetic glomerulosclerosis. Am J Cardiol. 1972 Nov 8;30(6):595-602. doi: 10.1016/0002-9149(72)90595-4. No abstract available. PMID 4263660
- [Result] Singh RM, Waqar T, Howarth FC, Adeghate E, Bidasee K, Singh J. Hyperglycemia-induced cardiac contractile dysfunction in the diabetic heart. Heart Fail Rev. 2018 Jan;23(1):37-54. doi: 10.1007/s10741-017-9663-y. PMID 29192360
- [Result] De Jong KA, Lopaschuk GD. Complex Energy Metabolic Changes in Heart Failure With Preserved Ejection Fraction and Heart Failure With Reduced Ejection Fraction. Can J Cardiol. 2017 Jul;33(7):860-871. doi: 10.1016/j.cjca.2017.03.009. Epub 2017 Mar 19. PMID 28579160
- [Result] Cook GA, Lavrentyev EN, Pham K, Park EA. Streptozotocin diabetes increases mRNA expression of ketogenic enzymes in the rat heart. Biochim Biophys Acta Gen Subj. 2017 Feb;1861(2):307-312. doi: 10.1016/j.bbagen.2016.11.012. Epub 2016 Nov 11. PMID 27845231
- [Result] Suhling K, Siegel J, Lanigan PM, Leveque-Fort S, Webb SE, Phillips D, Davis DM, French PM. Time-resolved fluorescence anisotropy imaging applied to live cells. Opt Lett. 2004 Mar 15;29(6):584-6. doi: 10.1364/ol.29.000584. PMID 15035478
- [Result] Wang M, Tang F, Pan X, Yao L, Wang X, Jing Y, Ma J, Wang G, Mi L. Rapid diagnosis and intraoperative margin assessment of human lung cancer with fluorescence lifetime imaging microscopy. BBA Clin. 2017 Apr 27;8:7-13. doi: 10.1016/j.bbacli.2017.04.002. eCollection 2017 Dec. PMID 28567338
- [Result] Luo T, Lu Y, Liu S, Lin D, Qu J. Phasor-FLIM as a Screening Tool for the Differential Diagnosis of Actinic Keratosis, Bowen's Disease, and Basal Cell Carcinoma. Anal Chem. 2017 Aug 1;89(15):8104-8111. doi: 10.1021/acs.analchem.7b01681. Epub 2017 Jul 18. PMID 28661125
- [Result] Jing Y, Wang Y, Wang X, Song C, Ma J, Xie Y, Fei Y, Zhang Q, Mi L. Label-free imaging and spectroscopy for early detection of cervical cancer. J Biophotonics. 2018 May;11(5):e201700245. doi: 10.1002/jbio.201700245. Epub 2018 Jan 30. PMID 29205885
- [Result] Farwell DG, Meier JD, Park J, Sun Y, Coffman H, Poirier B, Phipps J, Tinling S, Enepekides DJ, Marcu L. Time-resolved fluorescence spectroscopy as a diagnostic technique of oral carcinoma: Validation in the hamster buccal pouch model. Arch Otolaryngol Head Neck Surg. 2010 Feb;136(2):126-33. doi: 10.1001/archoto.2009.216. PMID 20157056
- [Result] Lagarto J, Dyer BT, Talbot C, Sikkel MB, Peters NS, French PM, Lyon AR, Dunsby C. Application of time-resolved autofluorescence to label-free in vivo optical mapping of changes in tissue matrix and metabolism associated with myocardial infarction and heart failure. Biomed Opt Express. 2015 Jan 7;6(2):324-46. doi: 10.1364/BOE.6.000324. eCollection 2015 Feb 1. PMID 25780727